CLINICAL TRIAL: NCT01935453
Title: A Phase I Study of Recombinant hGM-CSF Herpes Simplex Virus
Brief Title: A Phase I Study of Recombinant hGM-CSF Herpes Simplex Virus to Treat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OrienGene Biotechnology Ltd. (Industry)
Collaborators: START Shanghai (Unknown); Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OrienGene-01
Record Dates: First submitted 2013-08-23; First posted 2013-09-05 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2011-12

CONDITIONS: Melanoma; Liver Cancer; Pancreatic Cancer; Lung Cancer
MeSH Terms: conditions — Melanoma; Liver Neoplasms; Pancreatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant HSV-1 Injection (Experimental): Intratumoral injection Single dose: 4 groups -- 106 pfu, 107 pfu, 108 pfu and 4×108 pfu Multiple dose (three injections, every 2 weeks): 2 groups -- 108, 108, 108pfu and 4×108, 4×108, 4×108pfu Continuous treatment: Upon 4 weeks follow-up after administration, if the investigator deems that continuous treatment will benefit subjects, continuous intratumoral injection may be given, and the interval between each injection will be 2 weeks.
  Interventions: Biological: Recombinant hGM-CSF Herpes Simplex Virus Injection

INTERVENTIONS:
Biological: Recombinant hGM-CSF Herpes Simplex Virus Injection
  Other Names: OrienX010

SUMMARY:
The main purpose of this study is to study the safety of OrienX010 in the treatment of kinds of solid tumors such as melanoma,liver cancer,pancreatic cancer and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients in advanced stage of malignant tumor diagnosticated by pathologic and cytological analysis.
* lack of routine effective treatment,failure of routine treatment or relapse
* age of 18-70,ECOG 0-2 and estimated survival is above 3 months
* had an interval of above 4 weeks since exposure to chemotherapy or radiotherapy and above 6 weeks since exposure to nitrosoureas or mitomycin C.

Exclusion Criteria:

* Serious internal diseases
* uncontrolled primary and metastatic brain tumor
* sizes of tumor does not meet the requirement of injection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Exploring the MTD of OrienX010 according to DLT,which defined as the serious degree of adverse events relates to the medicine not less than grade 3 of CTCAE v4.03 | 28 days after the last administration

SECONDARY OUTCOMES:
Using RECIST 1.1 to evaluate the preliminary efficacy of OrienX010 | 28 days after the last administration

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Fudan University; Jun Ren, MD, Principal Investigator — Beijing Shijitan Hospital,CMU
Locations (2):
- China (2):
  - Beijing Shijitan Hospital,CMU, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality